CLINICAL TRIAL: NCT06889207
Title: Physical Exercise Prehabilitation Program in MEtabolic SuRgery
Acronym: PEPPER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Flevoziekenhuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL74088.018.20
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-10

CONDITIONS: Obesity and Overweight; Bariatric Surgery; Prehabilitation; Exercise; Physical Fitness; Six Minute Walk Test
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Preoperative Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prehabilitation (Active Comparator): Patients in the intervention group will have two supervised training sessions per week for eight weeks in group sessions supervised by a physiotherapist.
  Interventions: Behavioral: Physical exercise prehabilitation
- No prehabilitation (No Intervention): Receives no exercise prehabilitation program

INTERVENTIONS:
Behavioral: Physical exercise prehabilitation — Patients in the intervention group will have two supervised training sessions per week for eight weeks in group sessions supervised by a physiotherapist.
  Other Names: Prehabilitation; Exercise program
  Arms: Prehabilitation

SUMMARY:
The goal of this clinical trial is to learn if an exercise program before bariatric surgery works to treat obesity, could improve physical condition and weight loss before bariatric surgery and induce a lifestyle behavior change. The main questions it aims to answer are:

* Does a supervised exercise program lead to improved physical condition prior to bariatric surgery?
* Does a supervised exercise program prior to bariatric surgery lead to reduced surgery related complications?
* Does a supervised exercise program prior to bariatric surgery lead to maintained lifestyle changes after surgery?

Participants will:

* Receive either no training program or physical exercise training program twice a week, supervised by a physical therapist, for a duration of 8 weeks.
* Have their fitness measured at the start and at the end of the 8 weeks, measured with a six minute walking test.
* Fill in a survey on their perceived quality of life and exercise habits at the start of the trial, and at 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Body-Mass-Index (BMI) 40 kg/m2 or higher, or 35 kg/m2 or higher with the presence of at least one comorbidity (type 2 diabetes, high blood pressure, heart and/or vascular diseases, obstructive sleep apnea (OSA), dyslipidemia, or arthritis).
* Primary bariatric patients; without previous bariatric surgery. For inclusion the investigators will follow the National Guidelines on metabolic surgery.

Exclusion Criteria:

Patients with:

* mobility problems (patients who are not able to exercise)
* cognitive disabilities
* illiteracy (patients who are not able to read and understand the language of the country where the study will be performed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
six-minute walk test | 2 months
  Preoperative physical condition, assessed by using the six-minute walk test (6MWT). The target increase of the 6MWT is 10% in the intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- FlevoZiekenhuis, Almere Stad, Flevoland, Netherlands